CLINICAL TRIAL: NCT05986396
Title: Outcomes of Pulmonary Valve Replacement With the INSPIRIS (Model 11500A) Valve for Pulmonary Valve Replacement in Children and Young Adults
Brief Title: Outcomes of Pulmonary Valve Replacement With the INSPIRIS (Model 11500A) Valve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Victor Bautista Hernandez, Associate Professor of Surgery, Baylor College of Medicine
Other Study IDs: H-51357
Record Dates: First submitted 2023-07-12; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Heart Valve Prosthesis
Keywords: Pulmonary Valve Replacement; Pulmonary Valve; Congenital Heart Disease; INSPIRIS Resilia
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects: Subjects that have received the INSPIRIS Resilia device.
  Interventions: Device: INSPIRIS Resilia (model 11500A)

INTERVENTIONS:
Device: INSPIRIS Resilia (model 11500A) — Aortic Valve

SUMMARY:
The goal of this retrospective chart review is to contribute to the literature on the mid-term durability and hemodynamics of the INSPIRS Resilia bioprosthesis when implanted in children and young adults.

DETAILED DESCRIPTION:
The primary objective of our study is to contribute to the scarce body of literature on the mid-term durability and hemodynamics of the INSPIRIS Resilia (model 11500) bioprosthesis when implanted in the pulmonary position in children and young adults. Investigators also aim to identify: effect of age on SVD, freedom from SVD, pathology of SVD, valve-related complications, freedom from re-operation, and survival rate.

ELIGIBILITY:
Inclusion Criteria:

Subjects that have received the INSPIRIS Resilia device at participating institutions from 06/2017 through 12/2022.

Exclusion Criteria:

Subjects that have not received the INSPIRIS Resilia device.

Ages: 0 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with congenital heart disease that have received the INSPIRIS Resilia device.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Contribute to the scarce body of literature | 5 years after implantation
  The primary objective of our study is to contribute to the scarce body of literature on the mid-term durability and hemodynamics of the INSPIRIS Resilia (model 11500) bioprosthesis when implanted in the pulmonary position in children and young adults

SECONDARY OUTCOMES:
Identify the effect of age of the INSPIRIS Resilia (model 11500) bioprosthesis when implanted in the pulmonary position in children and young adults | 5 years after implantation
  Structural valve deterioration, freedom from SVD, valve related complications, freedom from re-operation, survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Victor Bautista-Hernandez, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine at CHRISTUS Children's, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No